CLINICAL TRIAL: NCT05996341
Title: The Effects of Blood Flow Restriction-based Abdominal draw-in Maneuver on Activation of Abdominal Core Muscles in Patients With Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH111-REC2-221
Record Dates: First submitted 2023-07-27; First posted 2023-08-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Non-specific Low Back Pain
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LBPADIM_BFR group (Experimental): Recipient No. 12 lower ribs and upper rechargeable nylon ribs , charge to 160mmHg and do ADIM at the same time and retract the abdominal muscles and let the belly fold inward and upward toward the spine and hold for 10 seconds, once.
  The total number of intervention was 20 minutes, once a time, a total of 4 minutes.
  Interventions: Device: blood flow restriction
- LBPADIM_shan BFR group (Placebo Comparator): The recipient has a rechargeable nylon rib under the 12th rib , but it is not filled and does not cause abdominal muscle BFR, which is used as the BFR of abdominal muscle.
  At the same time, we also do ADIM authentication,and retract the abdominal muscles and let the belly fold inward and upward toward the spine and hold for 10 seconds, once.
  The total number of intervention was 20 minutes, once a time, a total of 4 minutes.
  Interventions: Device: blood flow restriction
- HealthyADIM_BFR group (Experimental): Tested The top rechargeable nylon under the 12th rib , charge to 160mmHg and do ADIM password at the same time, and tand retract the abdominal muscles and let the belly fold inward and upward toward the spine and hold for 10 seconds, once.
  The total number of intervention was 20 minutes, once a time, a total of 4 minutes.
  Interventions: Device: blood flow restriction

INTERVENTIONS:
Device: blood flow restriction — 12 lower ribs and upper rechargeable nylon ribs (84 cm long, 14 cm long) Points), recharge to 160mmHg
  Other Names: Delfi's Personalized Tourniquet System

SUMMARY:
The transverse abdominis (TrA) is the deepest muscle layer of lateral and anterior abdominal wall and also known as a significant component of core stability. Abdominal draw-in maneuver (ADIM) is the main for the strengthening of the deep muscle, however, sufficient activation of TrA by ADIM is limited. Blood flow restriction (BFR) training is a technique combined with low intensity exercise that produces similar results to high intensity training. Therefore, the purpose of this study is to explore whether BFR-assisted ADIM can become a new auxiliary way to train TrA, and whether it can better activate their TrA in patients with low back pain. Low back pain (LBP) is a major health problem with huge economic and social costs. Core muscle weakness is a risk factor for LBP. Past studies have also pointed out that the biggest cause affecting the quality of life and activities of modern people is lower back pain. In modern life, low back pain can be said to be a very common disease. According to past research, there is a 50% to 70% chance that people may have lower back pain in their lifetime, and non-specific low back pain accounts for the majority (90%), the reason why the influence of non-specific low back pain is so great is not only physically but also psychologically. When people perform many functions of daily life, people need the help of the waist. But once the wrong way of effort or posture will lead to more pressure on the spine, leading to greater pain, a strong sense of discomfort will haunt them for a long time. Therefore, the activation and control of TrA is very important because of the relationship between the lateral direction of TrA, so when TrA contracts, it will result in a decrease in waist circumference, an increase in thoracolumbar fascia tension and an increase in intra-abdominal pressure, so it is regarded as the most important stable muscle in the core.In addition, TrA is a special presence in the core muscle group, it can independently contract and like the presence of waist protection to stabilize our spine, but because it is located in the deepest layer, coupled with less muscle activity, it is difficult to effectively activate correctly, so if TrA is not activated or contracted correctly, it may cause non-specific lower back pain.

DETAILED DESCRIPTION:
In this study, 20 healthy people and 20 patients with lower back pain were recruited and divided into healthy group, experimental group (patients with lower back pain) and sham experimental group (patients with lower back pain). The subjects in the experimental group and the healthy group were tied under the ribs with a pulse band (14 cm wide and 84 cm long) to block at least 60% of the blood flow and do abdominal exercise. In the sham experimental group, the ventral compression band was fastened but the abdominal contraction exercise was performed without inflation. Each subject exercised for 20 minutes twice a week for six weeks. At the first, third and sixth week, ultrasound (Ultrasound, USD) was used to evaluate the muscle thickness and muscle activation of external oblique muscle, internal oblique muscle and transverse muscle (core muscle group). This study expects that blood blocking training can increase the degree of activation, muscle strength and hypertrophy of transverse abdominal muscle in patients with lower back pain, and can provide a new auxiliary method to improve the predicament that it is difficult to activate transverse abdominal muscle correctly.

ELIGIBILITY:
Inclusion Criteria:

* Confirm that it is caused by pathological and mental stress or illness
* Non-idiopathic low back pain
* persistent or intermittent pain for more than six weeks
* the pain index of the scale, number is between 2 and 10 points.

Exclusion Criteria:

* Stress fracture
* osteoporosis
* acute lower back pain
* Spinal tumor
* spinal canal narrowing
* spinal osteitis
* spinal meningitis
* vertebral slippage

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | The experiment was conducted for a total of five weeks.After the first ultrasonic image estimation and the fourth week, all the assessments are carried out again, and then tracked down in the fifth week. Estimate.
  In this study, abdominal muscles were evaluated by Brightness-mode, 5M-Hz, Linear).
  The thickness of meat during abdominal muscle relaxation and during draw-in. The probing position is located at the lowest end of the rib and in the middle of the iliac spine.
  At the midpoint of the axillary line. Put an ultrasonic image of the abdominal muscle in the abdominal muscle and vomit in ADIM.
  At the end of the day, we take an image. Then calculate the muscle thickness. The calculation standard is from the tail and abdomen of TrA The fascia joint tip is three centimeters inward, and the muscle thickness of transvers abdominal, internal oblique and external oblique muscle is calculated from bottom to top, and Total muscle thickness, measured in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy of China Medical University, Taichung, Test2, Taiwan